CLINICAL TRIAL: NCT01018381
Title: Randomized Clinical Study of Arabinoxylan Rice Bran (MGN-3/Biobran) for the Treatment of Hepatocellular Carcinoma and Hepatitis B and C Infection
Brief Title: Arabinoxylan Rice Bran (MGN-3/Biobran) for the Treatment of Hepatocellular Carcinoma and Hepatitis B and C Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The 108 Military Central Hospital (Other Government)
Collaborators: Charles Drew University of Medicine and Science (Other)
Responsible Party: Mai Hong Bang, M.D. Ph.D., The 108 Military Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC and HBV
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B
Keywords: HCC; HBV; MGN-3; BioBran; Alternative Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — Radiofrequency Ablation; polysaccharide MGN3; lens intermediate filament proteins; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Therapy (Active Comparator): Conventional therapy is given, including PEIT, TOCE, PEIT + TOCE, TOCE + RFA for hepatocellular carcinoma or Entecavir for hepatitis B virus.
  Interventions: Procedure: PEIT; Procedure: TOCE; Procedure: TOCE plus PEIT; Procedure: TOCE plus RFA; Drug: Entecavir
- Conventional Therapy plus MGN-3 (Experimental)
  Interventions: Procedure: PEIT; Procedure: TOCE; Procedure: TOCE plus PEIT; Procedure: TOCE plus RFA; Dietary Supplement: MGN-3; Drug: Entecavir

INTERVENTIONS:
Procedure: PEIT — For patients with HCC: Ethanol (99.5%) 3-15 ml/treatment(mean 8ml/treatment) , 2 times/week (mean 6 treatment/patient). For patients with a tumor size under 5 cm in diameter, we applied the formula of M. Ebara: V = 4/3∏ (r+0.5)3 (V: total Ethanol volume, r: radius of tumor).
  Precise treatment was dependent on tumor size, outcomes after first PEIT treatment and time to recurrence of disease.
  Other Names: Pericutaneous Ethanol Injection Therapy; Pericutaneous Ethanol Injection; PEI
Procedure: TOCE — For patients with HCC: Adriamycine was mixed with lipiodol, Adriamycine 20-60mg/treatment (mean 40mg/treatment),lipiodol 5-20ml/treatment(mean 12ml/treatment), 1-2 months between treatments, 2-5 treatments/patient (mean 3 times/patient), which depended on tumor size, outcomes after first TOCE and time to recurrence of disease.
  Other Names: Transarterial oily chemoembolization
Procedure: TOCE plus PEIT — A combination of transarterial oily chemoembolization and pericutaneous ethanol injection therapy are given for patients with HCC.
  Other Names: Transarterial oily chemoembolization; Pericutaneous ethanol injection therapy; Pericutaneous ethanol injection
Procedure: TOCE plus RFA — For patients with HCC: A combination of transarterial oily chemoembolization plus radiofrequency ablation is given. For RFA: On mission 60w/s , 5minutes/circle, 2-4 circles/treatment, 1-2 treatments/week (tumor size under 2cm: 1 treatment; 2-4 cm: 2-3 treatments,over 4 cm: 3-5 treatments)
  Other Names: Transarterial oily chemoembolization; Radiofrequency ablation
Dietary Supplement: MGN-3 — For patients with HCC or hepatitis B, arabinoxylan rice bran food supplement is given. 1 gram per day, every day, for a duration of 12 months. For the MGN-3 group, the interventional therapy was given with MGN-3 simultaneously.
  Other Names: Peak Immune 4; BioBran; Lentin Plus 1000
  Arms: Conventional Therapy plus MGN-3
Drug: Entecavir — For patients with hepatitis B viral infection, a dose of 0.5mg/day, every day, was given for a duration of 24 months.
  Other Names: Baraclude

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common cancer worldwide with an estimated 626,000 new cases per year worldwide, accounting for 5.7% of new cancer cases. Although resection and transplantation offer the best 5-year survival rates, not all patients are suitable surgery candidates. Other treatments include pericutaneous ethanol injection (PEI), radiofrequency ablation (RFA), and transarterial oily chemoembolization (TOCE), all of which enhance the survival rate and aid in shrinkage of the tumor. The very low survival rate among HCC patients, 3-5%, reflects the inadequacy of conventional therapies for the disease and highlights the necessity of finding new treatments or modifying the current treatment.

The hepatitis B virus (HBV) causes liver disease that can range in severity from a mild illness that lasts several weeks (acute hepatitis B) to a long-term chronic illness. An estimated 2 billion people have been infected with HBV worldwide, resulting in more than 350 million individuals with chronic, long-term liver infections. Patients with chronic HBV infection are at a great risk for the development of cirrhosis, hepatic failure, and HCC. There is no cure for hepatitis B and care is mostly palliative. There are several anti-viral and interferon drugs, such as Entecavir and Interferon α therapy, which can help some patients. However, these drugs are costly, thousands of dollars per year, and are not widely available in many countries, especially in the developing world. Vaccination is available and effective and is recommended for all individuals at risk for HBV infection. However, vaccination is only effective in individuals who have not been exposed to HBV. Hepatitis B is closely linked to liver cancer, which is almost always fatal.

MGN-3/Biobran is an arabinoxylan extracted from rice bran that is treated enzymatically with an extract from Shiitake mushrooms. MGN-3 demonstrated anti-cancer activity in vivo in mice and humans. The present study was carried out to examine whether combining the current conventional treatment with a food supplement, arabinoxylan rice bran (MGN-3/Biobran), may improve the outcome of the disease and increase the survival rate of patients with HCC or HBV. We hypothesize that a combinatory treatment of conventional therapy with MGN-3/Biobran will augment the therapeutic effect seen when patients are treated with conventional therapy alone.

DETAILED DESCRIPTION:
Objective(s): The objective of this study is to analyze a data from a study that examined the biotherapeutic effect of combining conventional therapy in the presence of MGN-3/Biobran. The study focused on treatment of patients in Vietnam with hepatocellular carcinoma (HCC) and Hepatitis B and C.

Purpose of the study:

Aim 1: The biotherapeutic effect of combining conventional therapy and a natural, non-toxic arabinoxylan rice bran (MGN-3/Biobran) for the treatment of patients with HCC will be examined. Parameters under investigation include, lifespan of the patient, progression of the disease (tumor size), and recurrence of the disease.

Aim 2: The biotherapeutic effect of combining conventional therapy and a natural, non-toxic arabinoxylan rice bran (MGN-3/Biobran) for the treatment of patients with Hepatitis B virus (HBV) will be examined. Parameters under investigation include alanine transaminase (ALT) levels, HBV antigen levels, and HBV DNA levels.

Methodology:

Study Design:

Secondary analysis of data from "The effects of Biobran/Lentin Plus in the adjuvant therapy of hepatocellular carcinoma and chronic hepatitis B" study. The study was a randomized controlled design that was conducted from 6/2006 to 7/2008 at the 108 Military Central Hospital, Hanoi, Vietnam with Dr. Mai Hong Bang as the Principal Investigator. MGN-3/Biobran was approved by Vietnam Ministry of Health with import VISA No.12577/2005/CBCL-YT. Therefore, The 108 Military Central Hospital approved the study for treatment of patients with HCC and hepatitis B too.

1. Hepatocellular Carcinoma (HCC): Sixty-eight patients of both sexes, male and female, with HCC were divided into two groups: group 1 (38 patients) was treated with conventional therapy plus MGN-3 for 3 years, and group 2 (30 patients) was treated with conventional therapy alone. At various intervals and at the end of the study patients were assessed for the following: lifespan of the patient, progression of the disease (tumor size), and recurrence of the disease.
2. Hepatitis B virus (HBV): Sixty-two patients of both sexes, male and female, with HBV were divided into two groups: group 1 (32 patients) was treated with conventional therapy plus MGN-3 for 3 years, and group 2 (30 patients) was treated with conventional therapy alone. Conventional therapy given was the anti-viral drug, Entecavir.

   Data were collected every six months for two years. Parameters under investigation included: alanine transaminase (ALT) levels, HBV antigen (HeBAg), and HBV DNA levels.

   Patients were treated with standard treatment (transarterial oily chemoembolization (TOCE) for HCC; Entecavir for HBV) in combination with the experimental treatment, arabinoxylan rice bran (MGN-3/Biobran) and compared with a control group given standard treatment alone. Standard treatment was administered for 3 years. The experimental treatment (MGN-3/Biobran) was administered at a dose of 1g/day for 3 years.

   Patient characteristics and measures:
   * Group: two groups Group1 = Conventional therapy Group2 = Conventional therapy + MGN-3
   * Age range of the patients: 30-68 years old
   * Gender: male and female
   * Medical condition(s):

   Hepatitis infection:

   Hepatitis B: HCC HBV Hepatitis C: HCC Hepatitis B and C: HCC
   * Number of tumors/patient (HCC study)
   * Tumor size (HCC study): was measured in cm. <3 cm 3-6cm >6cm
   * AFP level: HCC - ≤500 ng/ml >500 ng/ml
   * HBV viral load
   * ALT level: HCC
   * HBV <100 IU/ml 100-250 IU/ml: 37 patients >250 IU/ml: 15 patients
   * Tumor Recurrence
   * Patient Survival

   Intervention details Treatment group(s): HCC - Intervention only (PEIT, TOCE, PEIT + TOCE, TOCE + RFA) Intervention + MGN-3 HBV - Intervention only (Entecavir) Intervention + MGN-3 Control(s): Intervention only group served as a control Co-interventions: Intervention + MGN-3 group Duration of intervention: HCC - 3 years HBV - 2 years

   Who delivered intervention? Dr. Mai Hong Bang and some other doctors. A consultation before delivering intervention for all patients

   Outcome measures HCC: ALT level, AFP level, tumor size, patient survival, recurrence HBV: ALT level, HBV DNA level, recurrence, patient survival, HBeAg seroconversion

   Methods of assessing outcome measures:

   ALT and AFP levels, HBV DNA level, HBeAg seroconversion: blood test Tumor size: ultrasonography and radiography Patient survival: observation

   When were they measured? Every 6 months Length of follow-up: HCC - 3 years HBV - 2 years

   Inclusion criteria:

   HCC patient Criteria of inclusion - Patient had ≤3 tumors (1 tumor under 12cm/ or 2 tumor under 5cm /or 3 tumor under 3cm) - Stage of disease: Okuda I,II and Child Pugh A,B
   * Liver biopsy: HCC positive
   * General condition: average/ good

   Chronic hepatitis B patient Criteria of inclusion

   - Patient have been carrying HBsAg over 6 months

   - ALT was over or equal 2 times ULN
   * HBV-DNA level: 104 (log10 copies/ml) with HBeAg(-) patient and 105 (log10 copies/ml) with HBeAg(+) patient

   Exclusion criteria:

   HCC patient Criteria of exclusion - Tumor size is too big (over 12 cm), multiple tumors (over 3 tumors or diffuse tumor type) - Prothrombin under 60%

   - Severe liver or/ and renal insufficiency
   * Portal vein body thrombosis

   Chronic hepatitis B patient Criteria of exclusion
   * Used immunotherapy or corticotherapy for 6 months
   * Pregnant woman

   Procedures: Upon approval by IRB, the data will be analyzed using statistical analysis and the data will be published in a peer-reviewed journal, as this data has not yet been published. We will receive the data from the PI (Dr. Mai Hong Bang, MD Ph.D., Associate Professor, Department of Hepatogastroenterology). After receiving the IRB approval, we will conduct secondary analysis of the data. We will receive the data as an electronic file excel file format with the code book for all the variables. We will do frequency and data checking and data management to prepare the data for analysis. We will do recoding and create new variables from the existed variables as a way to prepare for the data analysis.

   Benefits to subjects: Conventional therapies for HCC and HBV, in addition to their toxicity, do not substantially improve the survival rate of the patients. The combination of MGN-3/Biobran with these conventional therapies may improve the survival rate of the patients and decrease the rate of recurrence.

   Benefits to the Community: There is a disproportionately high incidence of HCC in developing countries, and over 50% of HCC cases occur in Asia. Hepatitis B is closely linked to liver cancer, which is almost always fatal. It is estimated that nearly 80% of all liver cancer worldwide is caused by hepatitis B infection. Therefore, there is a need for new treatments with minimal to no side effects to combat these diseases. This study will determine the potential of MGN-3/Biobran combined with conventional therapy to improve the outcome of these diseases.

ELIGIBILITY:
Inclusion criteria:

HCC patient Criteria of inclusion

* Patient had ≤3 tumors (1 tumor under 12cm/ or 2 tumor under 5cm /or 3 tumor under 3cm)
* Stage of disease: Okuda I,II and Child Pugh A,B
* Liver biopsy: HCC positive
* General condition: average/ good

Chronic hepatitis B patient Criteria of inclusion

* Patient have been carrying HBsAg over 6 months
* ALT was over or equal 2 times ULN
* HBV-DNA level: 104 (log10 copies/ml) with HBeAg(-) patient and 105 (log10 copies/ml) with HBeAg(+) patient

Exclusion criteria:

HCC patient Criteria of exclusion

* Tumor size is too big (over 12 cm), multiple tumors (over 3 tumors or diffuse tumor type)
* Prothrombin under 60%
* Severe liver or/ and renal insufficiency
* Portal vein body thrombosis

Chronic hepatitis B patient Criteria of exclusion

* Used immunotherapy or corticotherapy for 6 months
* Pregnant woman

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-06; Primary Completion 2008-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Patient survival | 3 years

SECONDARY OUTCOMES:
Disease recurrence | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mai Hong Bang, M.D. Ph.D., Principal Investigator — The 108 Military Central Hospital, Hanoi, Vietnam
Locations (1):
- The 108 Military Central Hospital, Hanoi, Vietnam